CLINICAL TRIAL: NCT05492851
Title: A Double-blind, Randomized Trial Comparing Three Single Dose Injections for Knee Osteoarthritis
Brief Title: Trial Comparing Three Single Dose Injections for Knee Osteoarthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study has only enrolled 6 subjects in 6 months since study initiation. Potential participants are unwilling to participate in the study due to the randomziation and blinding. Both aspects are needed to ensure a robust comparison between groups.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michael Baria, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022H0168
Record Dates: First submitted 2022-08-04; First posted 2022-08-09 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Triamcinolone; hylan; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Zilretta (Active Comparator): Generic Name: Triamcinolone acetonide Zilretta is an extended-release synthetic corticosteroid indicated as an intra-articular injection for the management ofosteoarthritis pain of the knee.
  5mL suspension of 32 mg of triamsinolone administered as a 1 dose parapatellar intra-articular injection.
  Interventions: Drug: Zilretta
- Synvisc One (Active Comparator): Generic Name: Hylan G-F 20 Synvisc-One combines the three doses of SYNVISC (hylan G-F 20) which consists of hylan A (average molecular weight6,000,000 daltons) and hylan B hydrated gel in a buffered physiological sodium chloride solution, pH 7.2.
  Each 10 mL syringe of Synvisc-One combines the three 2-mL doses (16 mg each) of a complete SYNVISC treatment regimen (48 mg). Synvisc-One belongs to a class of drugs called Intra-Articular Agents; Rheumatologics, Other.
  10mL of Hylan G-F 20 administered as a 1 dose parapatellar intra-articular injection.
  Interventions: Drug: Synvisc-One 48 MG in 6 ML Prefilled Syringe
- Monovisc (Active Comparator): Generic Name: Hyaluronan The Monovisc™ device is a proprietary high molecular weight hyaluronic acid (HA) viscosupplementation intended for the treatment of pain in patients with moderate osteoarthritis (OA) of the knee who have failed conservative non-pharmacological therapy and simple analgesics. The device is administered by a single injection via the para-patellar approach under sterile conditions.
  4mL injection of Hyaluronan administered as a 1 dose parapatellar intra-articular injection.
  Interventions: Drug: Monovisc 88 MG Per 4 ML Prefilled Syringe

INTERVENTIONS:
Drug: Zilretta — Intra-articular injection to treat knee osteoarthritis
  Arms: Zilretta
Drug: Synvisc-One 48 MG in 6 ML Prefilled Syringe — Intra-articular injection to treat knee osteoarthritis
  Arms: Synvisc One
Drug: Monovisc 88 MG Per 4 ML Prefilled Syringe — Intra-articular injection to treat knee osteoarthritis
  Arms: Monovisc

SUMMARY:
This study is a 3-arm, double-blind, randomized trial comparing the clinical outcomes of Zilretta, Synvisc One, and Monovisc for knee OA.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a leading cause of disability worldwide.1,2 Standard of care treatments for knee OA include activity modification, weight loss, therapeutic exercise and medications like non-steroidal anti-inflammatory drugs (NSAIDs). If these measures fail, injections like corticosteroids and hyaluronate (HA) can be helpful for pain control.3

The aforementioned injections have unique mechanisms of action. Steroid injections work through reducing joint inflammation, while HA works by lubricating and cushioning the joint. There are several varieties of steroids and HA injections that have been approved by the Food and Drug Administration for use in knee OA.

Among these variations are extended-release triamcinolone (Zilretta), hylan GF-20 (synvisc one), and hyaluronan (monovisc). While each are FDA approved and commonly used in orthopedic and sports medicine clinics, they have never been directly compared in any study. Therefore, when selecting a treatment for a patient, it is largely based on provider preference, not clinical data.

This study is a 3-arm, double-blind, randomized trial comparing the clinical outcomes of Zilretta, Synvisc One, and Monovisc for knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-85 years
* BMI < 40
* Diagnosis of unilateral knee OA
* Radiographic evidence of OA of the target knee (Kellgren-Lawrence grades 2-4)
* Continued OA pain in the target knee despite at least 6 weeks of: physical therapy and at least one of the following: activity modification (such as reducing impact on the knee), weight loss, and a 2 week trial of NSAID / acetaminophen.
* Knee Osteoarthritis Outcomes Score (KOOS)-Pain subscale 20-65
* Working knowledge of English language (to be able to complete all outcome scores)
* Ability to attend all follow-up appointments

Exclusion Criteria:

* 3+ effusion of the target knee (stroke test grading system)
* Prior injection therapy:

  * Steroid injection in target knee in the last 3 months
  * Viscosupplementation in target knee in the last 6 months
  * PRP in the target knee in the last 6 months
  * Cellular treatments in index knee (bone marrow, amniotic suspensions etc) 1 year
  * Participation in any experimental device or drug study within 1 year before screening visit
* Oral or IM steroids in the last 3 months (Inhaled steroids used in the treatment of asthma/allergies are permitted)
* Medical condition that may impact outcomes of procedure including:

  * Systemic inflammatory disorders that impact the joints like rheumatoid arthritis, lupus, etc
  * Undergoing current cancer treatment (other than non-melanoma skin malignancies)
* Taking immunosuppressants
* Previous cartilage repair procedure on the injured cartilage surface (ie, OATS, ACI, MFX) in the last 5 years
* Previous surgery at the target knee within the past 1 year
* Any degree of cognitive impairment
* Symptomatic OA of any other joint in the lower limbs
* Pregnancy, lactating, or intent to become pregnant during treatment period (Female participants will be asked if they are pregnant, lactating, or intend to become pregnant during treatment)
* Gout, Pseudogout (including radiographic evidence of chondrocalcinosis)
* History of infection or current infection at the affected joint
* Smoking (Former smokers< 1 year from quit date)

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) Pain patient reported outcome questionnaire | 6 month
  KOOS Pain evaluates short-term and long-term pain in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee pain.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) Symptoms patient reported outcome | Baseline, 3 month, 6 month
  KOOS symptoms evaluates short-term and long-term symptoms in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee symptoms.
Knee injury and Osteoarthritis Outcome Score (KOOS) Function in daily living (ADL) patient reported outcome | Baseline, 3 month, 6 month
  KOOS ADL evaluates short-term and long-term function in daily living in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee related issues in regards to daily living activity.
Knee injury and Osteoarthritis Outcome Score (KOOS) Function in Sport and Recreation (Sport/Rec) patient reported outcome | Baseline, 3 month, 6 month
  KOOS Sport/Rec evaluates short-term and long-term function in sports and recreation in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee related issues in regards to sports or recreation activity.
Knee injury and Osteoarthritis Outcome Score (KOOS) knee related quality of life (QOL) patient reported outcome | Baseline, 3 month, 6 month
  KOOS QOL evaluates short-term and long-term knee quality of life in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee related issues in regards to quality of life.
Knee injury and Osteoarthritis Outcome Score (KOOS) Pain patient reported outcome | Baseline, 3 month
  KOOS Pain evaluates short-term and long-term pain in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee pain.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baria, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Jameson Crane Sports Medicine Institute, Columbus, Ohio
  - Ohio State Outpatient Lewis Center, Lewis Center, Ohio

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared.